CLINICAL TRIAL: NCT01297335
Title: Hemodynamic Effect of Intrathecal Clonidine in Hypertensive Subjects: A Pilot Study to Assess Its Effectiveness in Hypertensive Subjects With Poor Blood Pressure Control (Phase II)
Brief Title: Effect of Intrathecal Clonidine in Hypertensive Subjects With Poorly Controlled Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Center for Clinical Research, Winston-Salem, NC (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1461 Clonidine; 1461 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: intrathecal; clonidine; poorly; controlled; hypertension
MeSH Terms: conditions — Hypertension | interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrathecal Clonidine (Experimental): Subject will receive one time Clonidine injection via lower lumber interspace. Clonidine (Duraclon), 100 μg/ml, 1.5 ml will be diluted to 2 ml with preservative free saline, and total of 150 μg will be delivered. Supine and sitting blood pressures and heart rate will be measured at 10 minute intervals until 60 minutes after clonidine administration, then at 15 minutes for next 3 hours.
  Interventions: Drug: clonidine

INTERVENTIONS:
Drug: clonidine — Intrathecal Clonidine
  Other Names: catapres

SUMMARY:
The purpose of this study is to determine the acute efficacy of intrathecal clonidine to reduce blood pressure in hypertensive subjects with poor blood pressure control and describe its effects on cardiovascular function.

DETAILED DESCRIPTION:
Hypertension occurs commonly, is associated with major morbidity and mortality, and responds poorly to current therapies in a small minority of compliant patients. The goal of this investigator-initiated study is to determine whether intrathecal administration of clonidine reduces blood pressure in hypertensive patients, focusing on a group who often achieve inadequate blood pressure control with multiple drug therapy.

After consent, pts will be screened and if qualified brought into center and intrathecal injection of clonidine given. Patients will be closely monitored for 4 hours, while data is collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hypertension
* Stable systolic blood pressure >140 mmHg and < 190 mmHg
* On 3 or more antihypertensive medications
* On a diuretic
* Patients must be able to understand the risks

Exclusion Criteria:

* Allergy to clonidine
* Presently on clonidine orally or transdermally
* Known or suspected correctable causes of secondary hypertension
* Breast Feeding or Pregnant women
* Unstable Ischemic Heart Disease
* Unstable Angina
* Intracoronary Stent Placement
* Coronary bypass within last 6 months
* Myocardial Infarction within last 6 months
* Congestive Failure
* Cardiac Arrhythmias
* Known Cerebral Vascular Disease
* Renal Disease
* Evidence of Injection Site Infection
* Known Bleeding Disorders
* Hepatic Insufficiency
* Renal Insufficiency
* Participation in an investigational drug study within 30 day of enrollment
* Prohibited Medications:

  * Clonidine
  * Yohimbine
  * Tricyclic Antidepressants
  * Mirtazapine
  * Digitalis
  * Reserpine
  * Guanethidine
  * Non-Steroidal Anti-inflammatory Medication
  * Alcohol or Barbiturates within 48 hours of study procedure

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. Rauck, MD, Principal Investigator — Owner

IPD SHARING:
Plan to Share IPD: No
no individual's data will be shared with anyone other than the members of the study staff, and the confidentiality will be maintained in accordance with HIPAA rules.

REFERENCES:
- [Background] Onesti G, Schwartz AB, Kim KE, Swartz C, Brest AN. Pharmacodynamic effects of a new antihypertensive drug, Catapres (ST-155). Circulation. 1969 Feb;39(2):219-28. doi: 10.1161/01.cir.39.2.219. No abstract available. PMID 4884576
- [Background] Davies DS, Wing AM, Reid JL, Neill DM, Tippett P, Dollery CT. Pharmacokinetics and concentration-effect relationships of intervenous and oral clonidine. Clin Pharmacol Ther. 1977 May;21(5):593-601. doi: 10.1002/cpt1977215593. PMID 870272
- [Background] Frisk-Holmberg M, Paalzow L, Wibell L. Relationship between the cardiovascular effects and steady-state kinetics of clonidine in hypertension. Demonstration of a therapeutic window in man. Eur J Clin Pharmacol. 1984;26(3):309-13. doi: 10.1007/BF00548760. PMID 6734692
- [Background] Reid JL, Wing LM, Mathias CJ, Frankel HL, Neill E. The central hypotensive effect of clonidine. Studies in tetraplegic subjects. Clin Pharmacol Ther. 1977 Apr;21(4):375-81. doi: 10.1002/cpt1977214375. PMID 321174
- [Background] Brown MJ, Struthers AD, di Silvio L. Peripheral alpha 2 adrenoceptor stimulation contributes to the sympatholytic effect of guanfacine in humans. J Cardiovasc Pharmacol. 1985;7 Suppl 6:S159-61. doi: 10.1097/00005344-198500076-00027. PMID 2414580
- [Background] Guthrie GP Jr, Kotchen TA. Effects of prazosin and clonidine on sympathetic and baroreflex function in patients with essential hypertension. J Clin Pharmacol. 1983 Aug-Sep;23(8-9):348-54. doi: 10.1002/j.1552-4604.1983.tb02747.x. PMID 6630584
- [Background] Mohanty PK, Sowers JR, McNamara C, Thames MD. Reflex vasoconstrictor responses to cardiopulmonary baroreceptor unloading, head-up tilt, and cold pressor testing in elderly mild-to-moderate hypertensives: effect of clonidine. J Cardiovasc Pharmacol. 1987;10 Suppl 12:S135-7. PMID 2455165
- [Background] Muzi M, Goff DR, Kampine JP, Roerig DL, Ebert TJ. Clonidine reduces sympathetic activity but maintains baroreflex responses in normotensive humans. Anesthesiology. 1992 Nov;77(5):864-71. doi: 10.1097/00000542-199211000-00005. PMID 1443738
- [Background] Houston MC. Treatment of hypertensive emergencies and urgencies with oral clonidine loading and titration. A review. Arch Intern Med. 1986 Mar;146(3):586-9. PMID 3513726
- [Background] Masotti G, Scarti L, Poggesi L, Bisi G, Gallini C, Neri Serneri GG. Changes in cardiac function after effective treatment of hypertensive emergencies with i.v. clonidine. Eur Heart J. 1984 Dec;5(12):1036-42. doi: 10.1093/oxfordjournals.eurheartj.a061605. PMID 6534750
- [Background] Niarchos AP. Evaluation of intravenous clonidine in hypertensive emergencies. J Clin Pharmacol. 1978 Apr;18(4):220-8. doi: 10.1002/j.1552-4604.1978.tb01596.x. PMID 632367
- [Background] Magorien RD, Hermiller JB, Unverferth DV, Leier CV. Regional hemodynamic effects of clonidine in congestive heart failure. J Cardiovasc Pharmacol. 1985 Jan-Feb;7(1):91-6. doi: 10.1097/00005344-198501000-00015. PMID 2580157
- [Background] Zochowski RJ, Lada W. Intravenous clonidine treatment in acute myocardial infarction (with comparison to a nitroglycerin-treated and control group). J Cardiovasc Pharmacol. 1986;8 Suppl 3:S41-5. PMID 2429112
- [Background] Wallace AW, Galindez D, Salahieh A, Layug EL, Lazo EA, Haratonik KA, Boisvert DM, Kardatzke D. Effect of clonidine on cardiovascular morbidity and mortality after noncardiac surgery. Anesthesiology. 2004 Aug;101(2):284-93. doi: 10.1097/00000542-200408000-00007. PMID 15277909
- [Background] Byrd BF 3rd, Collins HW, Primm RK. Risk factors for severe bradycardia during oral clonidine therapy for hypertension. Arch Intern Med. 1988 Mar;148(3):729-33. PMID 3341873
- [Background] Kibler LE, Gazes PC. Effect of clonidine on atrioventricular conduction. JAMA. 1977 Oct 31;238(18):1930-2. PMID 578552
- [Background] Toussaint C, Cave D, Saoudi N, Moore N, Letac B. Electrophysiological effects of intravenous clonidine on sinus node function and conduction in man. J Cardiovasc Pharmacol. 1984 Jan-Feb;6(1):56-60. PMID 6199612
- [Background] Clementy J, Castagne D, Wicker P, Dallocchio M, Bricaud H. Study of the electrophysiologic properties of clonidine administered intravenously. J Cardiovasc Pharmacol. 1986;8 Suppl 3:S24-9. doi: 10.1097/00005344-198608003-00007. PMID 2429109
- [Background] Rupp H, Maisch B, Brilla CG. Drug withdrawal and rebound hypertension: differential action of the central antihypertensive drugs moxonidine and clonidine. Cardiovasc Drugs Ther. 1996 Jun;10 Suppl 1:251-62. doi: 10.1007/BF00120495. PMID 8827948
- [Background] Fuxe K, Tinner B, Bjelke B, Agnati LF, Verhofstad A, Steinbusch HG, Goldstein M, Hersh L, Kalia M. Monoaminergic and Peptidergic Innervation of the Intermedio-Lateral Horn of the Spinal Cord. Eur J Neurosci. 1990;2(5):451-460. doi: 10.1111/j.1460-9568.1990.tb00436.x. PMID 12106031
- [Background] Fuxe K, Tinner B, Bjelke B, Agnati LF, Verhofstad A, Steinbusch HG, Goldstein M, Kalia M. Monoaminergic and Peptidergic Innervation of the Intermedio-Lateral Horn of the Spinal Cord. Eur J Neurosci. 1990;2(5):430-450. doi: 10.1111/j.1460-9568.1990.tb00435.x. PMID 12106030
- [Background] Unnerstall JR, Kopajtic TA, Kuhar MJ. Distribution of alpha 2 agonist binding sites in the rat and human central nervous system: analysis of some functional, anatomic correlates of the pharmacologic effects of clonidine and related adrenergic agents. Brain Res. 1984 Mar;319(1):69-101. doi: 10.1016/0165-0173(84)90030-4. PMID 6324960
- [Background] Guyenet PG, Cabot JB. Inhibition of sympathetic preganglionic neurons by catecholamines and clonidine: mediation by an alpha-adrenergic receptor. J Neurosci. 1981 Aug;1(8):908-17. doi: 10.1523/JNEUROSCI.01-08-00908.1981. PMID 6286903
- [Background] Stevens CW, Yaksh TL. Time course characteristics of tolerance development to continuously infused antinociceptive agents in rat spinal cord. J Pharmacol Exp Ther. 1989 Oct;251(1):216-23. PMID 2795458
- [Background] Eisenach JC, Tong CY. Site of hemodynamic effects of intrathecal alpha 2-adrenergic agonists. Anesthesiology. 1991 Apr;74(4):766-71. doi: 10.1097/00000542-199104000-00021. PMID 1672580
- [Background] De Kock M. Site of hemodynamic effects of alpha 2-adrenergic agonists. Anesthesiology. 1991 Oct;75(4):715-6. doi: 10.1097/00000542-199110000-00046. No abstract available. PMID 1928792
- [Background] Eisenach JC, Hood DD, Curry R. Intrathecal, but not intravenous, clonidine reduces experimental thermal or capsaicin-induced pain and hyperalgesia in normal volunteers. Anesth Analg. 1998 Sep;87(3):591-6. doi: 10.1097/00000539-199809000-00018. PMID 9728835
- [Background] Kooner JS, Birch R, Frankel HL, Peart WS, Mathias CJ. Hemodynamic and neurohormonal effects of clonidine in patients with preganglionic and postganglionic sympathetic lesions. Evidence for a central sympatholytic action. Circulation. 1991 Jul;84(1):75-83. doi: 10.1161/01.cir.84.1.75. PMID 2060125
- [Background] Castro MI, Eisenach JC. Pharmacokinetics and dynamics of intravenous, intrathecal, and epidural clonidine in sheep. Anesthesiology. 1989 Sep;71(3):418-25. doi: 10.1097/00000542-198909000-00018. PMID 2774269
- [Background] Eisenach JC, Lysak SZ, Viscomi CM. Epidural clonidine analgesia following surgery: phase I. Anesthesiology. 1989 Nov;71(5):640-6. doi: 10.1097/00000542-198911000-00003. PMID 2817456
- [Background] Mendez R, Eisenach JC, Kashtan K. Epidural clonidine analgesia after cesarean section. Anesthesiology. 1990 Nov;73(5):848-52. doi: 10.1097/00000542-199011000-00009. PMID 2240674
- [Background] Huntoon M, Eisenach JC, Boese P. Epidural clonidine after cesarean section. Appropriate dose and effect of prior local anesthetic. Anesthesiology. 1992 Feb;76(2):187-93. doi: 10.1097/00000542-199202000-00005. PMID 1736694
- [Background] Eisenach JC, D'Angelo R, Taylor C, Hood DD. An isobolographic study of epidural clonidine and fentanyl after cesarean section. Anesth Analg. 1994 Aug;79(2):285-90. doi: 10.1213/00000539-199408000-00014. PMID 7639365
- [Background] Chiari A, Lorber C, Eisenach JC, Wildling E, Krenn C, Zavrsky A, Kainz C, Germann P, Klimscha W. Analgesic and hemodynamic effects of intrathecal clonidine as the sole analgesic agent during first stage of labor: a dose-response study. Anesthesiology. 1999 Aug;91(2):388-96. doi: 10.1097/00000542-199908000-00012. PMID 10443601
- [Background] D'Angelo R, Evans E, Dean LA, Gaver R, Eisenach JC. Spinal clonidine prolongs labor analgesia from spinal sufentanil and bupivacaine. Anesth Analg. 1999 Mar;88(3):573-6. doi: 10.1097/00000539-199903000-00020. PMID 10072008
- [Background] Rauck RL, Eisenach JC, Jackson K, Young LD, Southern J. Epidural clonidine treatment for refractory reflex sympathetic dystrophy. Anesthesiology. 1993 Dec;79(6):1163-9; discussion 27A. PMID 8267190
- [Background] Eisenach JC, Rauck RL, Buzzanell C, Lysak SZ. Epidural clonidine analgesia for intractable cancer pain: phase I. Anesthesiology. 1989 Nov;71(5):647-52. doi: 10.1097/00000542-198911000-00004. PMID 2817457
- [Background] Eisenach JC, DuPen S, Dubois M, Miguel R, Allin D; Epidural Clonidine Study Group. Epidural clonidine analgesia for intractable cancer pain. The Epidural Clonidine Study Group. Pain. 1995 Jun;61(3):391-399. doi: 10.1016/0304-3959(94)00209-W. PMID 7478682
- [Background] Eisenach J, Detweiler D, Hood D. Hemodynamic and analgesic actions of epidurally administered clonidine. Anesthesiology. 1993 Feb;78(2):277-87. doi: 10.1097/00000542-199302000-00011. PMID 8439023
- [Background] Eisenach JC, Hood DD, Tuttle R, Shafer S, Smith T, Tong C. Computer-controlled epidural infusion to targeted cerebrospinal fluid concentrations in humans. Clonidine. Anesthesiology. 1995 Jul;83(1):33-47. doi: 10.1097/00000542-199507000-00005. PMID 7605017
- [Background] Hood DD, Mallak KA, Eisenach JC, Tong C. Interaction between intrathecal neostigmine and epidural clonidine in human volunteers. Anesthesiology. 1996 Aug;85(2):315-25. doi: 10.1097/00000542-199608000-00013. PMID 8712447
- [Background] De Kock M, Eisenach J, Tong C, Schmitz AL, Scholtes JL. Analgesic doses of intrathecal but not intravenous clonidine increase acetylcholine in cerebrospinal fluid in humans. Anesth Analg. 1997 Apr;84(4):800-3. doi: 10.1097/00000539-199704000-00019. PMID 9085961
- [Background] Eisenach JC, Hood DD, Curry R. Relative potency of epidural to intrathecal clonidine differs between acute thermal pain and capsaicin-induced allodynia. Pain. 2000 Jan;84(1):57-64. doi: 10.1016/S0304-3959(99)00181-5. PMID 10601673
- [Background] Eisenach JC, De Kock M, Klimscha W. alpha(2)-adrenergic agonists for regional anesthesia. A clinical review of clonidine (1984-1995). Anesthesiology. 1996 Sep;85(3):655-74. doi: 10.1097/00000542-199609000-00026. No abstract available. PMID 8853097
- [Background] Baker A, Klimscha W, Eisenach JC, Li XH, Wildling E, Menth-Chiari WA, Chiari AI. Intrathecal clonidine for postoperative analgesia in elderly patients: the influence of baricity on hemodynamic and analgesic effects. Anesth Analg. 2004 Jul;99(1):128-134. doi: 10.1213/01.ANE.0000114549.17864.36. PMID 15281518
- [Background] Nishikawa T, Kimura T, Taguchi N, Dohi S. Oral clonidine preanesthetic medication augments the pressor responses to intravenous ephedrine in awake or anesthetized patients. Anesthesiology. 1991 Apr;74(4):705-10. doi: 10.1097/00000542-199104000-00014. PMID 2008952
- [Background] Wing LM, Reid JL, Davies DS, Neill EA, Tippett P, Dollery CT. Pharmacokinetic and concentration-effect relationships of clonidine in essential hypertension. Eur J Clin Pharmacol. 1977 Dec 28;12(6):463-9. doi: 10.1007/BF00561067. PMID 598422
- [Background] Abdelhammed AI, Smith RD, Levy P, Smits GJ, Ferrario CM. Noninvasive hemodynamic profiles in hypertensive subjects. Am J Hypertens. 2005 Feb;18(2 Pt 2):51S-59S. doi: 10.1016/j.amjhyper.2004.11.043. PMID 15752933
- [Background] Ferrario CM. New approaches to hypertension management: always reasonable but now necessary. Am J Hypertens. 2005 Feb;18(2 Pt 2):23S-25S. doi: 10.1016/j.amjhyper.2004.11.042. No abstract available. PMID 15752930
- [Background] Adji A, O'Rourke MF. Determination of central aortic systolic and pulse pressure from the radial artery pressure waveform. Blood Press Monit. 2004 Jun;9(3):115-21. doi: 10.1097/01.mbp.0000132426.32886.e0. PMID 15199304
- [Background] Lemogoum D, Flores G, Van den Abeele W, Ciarka A, Leeman M, Degaute JP, van de Borne P, Van Bortel L. Validity of pulse pressure and augmentation index as surrogate measures of arterial stiffness during beta-adrenergic stimulation. J Hypertens. 2004 Mar;22(3):511-7. doi: 10.1097/00004872-200403000-00013. PMID 15076156
- [Background] al'Absi M, Devereux RB, Lewis CE, Kitzman DW, Rao DC, Hopkins P, Markovitz J, Arnett DK. Blood pressure responses to acute stress and left ventricular mass (The Hypertension Genetic Epidemiology Network Study). Am J Cardiol. 2002 Mar 1;89(5):536-40. doi: 10.1016/s0002-9149(01)02305-0. PMID 11867037
- [Background] Hood DD, Eisenach JC, Tong C, Tommasi E, Yaksh TL. Cardiorespiratory and spinal cord blood flow effects of intrathecal neostigmine methylsulfate, clonidine, and their combination in sheep. Anesthesiology. 1995 Feb;82(2):428-35. doi: 10.1097/00000542-199502000-00013. PMID 7856901
- [Background] Yaksh TL, Rathbun M, Jage J, Mirzai T, Grafe M, Hiles RA. Pharmacology and toxicology of chronically infused epidural clonidine.HCl in dogs. Fundam Appl Toxicol. 1994 Oct;23(3):319-35. doi: 10.1006/faat.1994.1112. PMID 7835532

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intrathecal Clonidine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intrathecal Clonidine: All subjects met all inclusion and exclusionary criteria, and we report study subjects' demographic information in following sections.
Arm/Group | Intrathecal Clonidine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  African American, Non-hispanic | 7
  White, Non-hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 10
Duration of Hypertension Diagnosis [Mean (Full Range); unit: years] | 17 [6 to 25]
Number of active antihypertensive medications [Number; unit: participants]
  4 active antihypertensive medications | 8
  3 active antihypertensive medications | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure After Intrathecal Injection of Clonidine.
Description: Subjects baseline blood pressure (systolic blood pressure (SBP), and diastolic blood pressure (DBP)), and blood pressures after clonidine injection was compared against baseline to assess efficacy of clonidine in refractory hypertensive subjects. Subject's blood pressure was monitored continuously after intrathecal injection of clonidine until subjects blood pressure nadir and return to pre clonidine injection level. The mean value reported below are the average changes in blood pressure from baseline (pre clonidine injection) in both SBP and DBP during post clonidine injection blood pressure monitoring for 4 hours.
  Blood pressure measurements were collected every 10 minutes for first hour after injection, and every 15 minutes after the first hour, up to 4 hours were averaged to report the change from baseline.
Time Frame: Baseline, Every 10 Minutes for first hour after clonidine injection, and every 15 minutes after first hour, until 4 hours after clonidine injection
Population: All subjects met inclusion and exclusionary criteria, and was given an intrathecal injection of clonidine. They were followed for changes in blood pressure for 4 hours.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Intrathecal Clonidine: Subject received one time Clonidine injection via lower lumber interspace. Clonidine (Duraclon), 100 μg/ml, 1.5 ml will be diluted to 2 ml with preservative free saline, and total of 150 μg were delivered. Supine and sitting blood pressures and heart rate were measured at 10 minute intervals until 60 minutes after clonidine administration, then at 15 minutes for next 3 hours.
Arm/Group | Intrathecal Clonidine
Number analyzed (Participants) | 10
mm Hg
  Change in mean SBP after clonidine injection | 79 (28)
  Change in DBP after clonidine injection | 37 (17)

2. Secondary Outcome: Likert Scale Pain Rating
Description: Likert scale is 11 point digital pain rating system that asks subjects to rate their pain from 0 to 10. Rating of 0 means no pain at all, and in increasing order, 10 would mean worst pain imaginable/ unbearable pain.
Time Frame: Pre-dose and 1 hour post injection.
Population: All subjects met inclusion and exclusionary criteria, and received intrathecal injection of clonidine. Subjects were asked to rate their baseline pain on Likert scale prior to receiving intrathecal clonidine injection, and 1 hour post intrathecal clonidine injection.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intrathecal Clonidine
Number analyzed (Participants) | 10
units on a scale
  Pre-injection average Likert score | 6.5 (1.9)
  Post-injection average Likert score | 3.6 (2.6)

3. Secondary Outcome: Changes in Visual Analogue Scale (VAS) Ratings of Sedation and Sensation of Dry Mouth Reported by the Subjects, Pre and 1 Hour Post Injection
Description: Subjects were asked to rate severity of two of the most common side effects of clonidine, sedation and sensation of dry mouth, at pre and post (1 hour after) intrathecal administration of clonidine. The mean changes between pre and post injection VAS ratings of sedation and sensation of dry mouth are reported below. The VAS scale ranges from 1 to 10 cm, with higher values indicating higher level of sedation and higher level of dry mouth.
Time Frame: Before clonidine injection (Baseline), and at 1 hour after clonidine injection.
Population: All qualified subjects were given intrathecal clonidine and were asked to rate level of sedation and sensation of dry mouth before clonidine injection (baseline) and 1 hour post injection on VAS scale.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Intrathecal Clonidine: Subjects were asked to rate both level of sedation and dryness of their mouths (two of the most common side effects of clonidine) at before clonidine injection (baseline) and at one hour after clonidine injection (Post injection) on VAS scale. VAS scale is an analogue scale that measures subject response from 0 to 10 cm, where larger value represents greater level of sedation and dryness in the mouth subject experienced.
Arm/Group | Intrathecal Clonidine
Number analyzed (Participants) | 10
cm
  Change in level of sedation | 3.36 (3.66)
  Change in sensation of dry mouth | 3.47 (3.93)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the duration of the study. Some adverse events, such as pregnancy that occurred during the study would have been followed until the delivery of fetus or termination of pregnancy.
Description: Events such as spinal headaches, or hypotension requiring intravenous fluids or vasopressor intervention
Arm/Group | Intrathecal Clonidine
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
This study was limited by small sample size, and lack of control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No